CLINICAL TRIAL: NCT03430284
Title: Effects of Multifactorial Intervention on Type 2 Diabetes - A Multicenter, Open-Label, Randomized, Parallel Controlled, Community Trial.
Brief Title: Multifactorial Intervention on Diabetes (MIDiab Study)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shandong Provincial Hospital (Other Government)
Collaborators: The Affiliated Hospital of Qingdao University (Other); The First Hospital of Jilin University (Other); The First People's Hospital of Yinchuan (Other); Beijing Hospital, National Center of Gerontology (Unknown); The First Affiliated Hospital of Air Force Medicial University (Other); Inner Mongolia People's Hospital (Other); The Affiliated Hospital of Inner Mongolia Medical University (Other); Fujian Medical University Union Hospital (Other); The Fourth Affiliated Hospital of Harbin Medical University (Other); Yantai Yuhuangding Hospital Affiliated to Qingdao University (Unknown)
Responsible Party: Principal Investigator, Jia-jun Zhao, Professor, Shandong Provincial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017YFC1309800
Record Dates: First submitted 2018-01-22; First posted 2018-02-12 (Actual); Last update posted 2021-07-09 (Actual); Status verified 2021-07

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Type 2 Diabetes Mellitus; Diabetic Vascular Complications; Multifactorial Intervention; Digital and Network Management
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetic Angiopathies | interventions — Drug Therapy; Therapeutics

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Integrated Treatment (Experimental)
  Interventions: Behavioral: Lifestyle therapy; Drug: Pharmacotherapy; Other: Monitoring and management
- General Treatment (Other)
  Interventions: Other: General treatment

INTERVENTIONS:
Behavioral: Lifestyle therapy — The key components of lifestyle therapy include medical nutrition therapy, regular physical activity, sufficient amounts of sleep, behavioral support, and smoking cessation and avoidance of all tobacco products.
  Arms: Integrated Treatment
Drug: Pharmacotherapy — Pharmacological therapy is individualized. 1.Glucose-lowering agents:
  1. Oral antihyperglycemic agents:Biguanides;Sulfonylureas;Thiazolidinediones;Glinides;a-Glucosidase inhibitors;DPP-4 inhibitors;Sodium-glucose cotransporter 2 inhibitors
  2. GLP-1 receptor agonist
  3. Insulin:Rapid-acting analogs;Short-acting analogs;Intermediate-acting analogs;Basal insulin analogs;Premixed insulin products
  2.Blood pressure-lowering agents
  (1)ACE inhibitor;(2)Angiotensin receptor blockers (ARBs);(3)Calcium channel blockers (CCB);(4)Diuretics;(5)β-blockers;(6)α1-blockers
  3.Lipid-modifying agents
  (1)Statins;(2)Fibrates;(3)Others: Nicotinic Acid, Ezetimibe,Probucol,Bile Acid Sequestrants,Policosanol,etc.
  4.Medications for weight management
  (1)Glucose-lowering agents associated with weight loss;(2)Orlistat;(3)Metabolic Surgery
  The above medications are individualized to maintain the risk factors (blood glucose, serum lipid profiles, blood pressure and weight) at appropriate levels.
  Arms: Integrated Treatment
Other: Monitoring and management — Before follow-up, patients are divided into low, moderate or high risk for diabetic vascular complications. During follow-up, frequencies of interview and risk factor monitoring are formulated based on the risk stratification.
  Arms: Integrated Treatment
Other: General treatment — General treatment is carried out based on the device from the general practitioners at present.
  Arms: General Treatment

SUMMARY:
The prevalence of diabetes mellitus has been increasing in recent decades in China, and vascular complication is the major burden in patients with type 2 diabetes. Previous studies demonstrated that only glycemic control was not effective enough to prevent or improve diabetic vascular complications, but guidelines from the Chinese Diabetes Society and other national guidelines recommend an integrated multifactorial treatment approach. In this study, we aim to evaluate the effect on diabetic vascular complications of a multifactorial intervention comprising behavior modification, polypharmacological therapy and periodical monitoring in patients with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

1. 35-75 years old;
2. diagnosed as type 2 diabetes according to the criteria of the World Health Organization in 1999.

Exclusion Criteria:

1. type 1 diabetes，specific types of diabetes，gestational diabetes or pregestational diabetes;
2. acute cardiovascular or cerebrovascular accidents within past 3 months;
3. severe hepatic or renal dysfunction;
4. malignant tumor;
5. allergic history or contraindication for any drugs in trials;
6. taking part in other clinical trials;
7. obviously poor compliance.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6300 (Estimated)
Dates: Start 2018-04-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Integrated management rate of multiple risk factor in type 2 diabetes | 30 months
  Multiple risk factor: plasma glucose, blood pressure, serum lipid profiles and obesity
Incidence of diabetic vascular complications | 30 months
  Diabetic vascular complications: both macrovascular and microvascular complications
Control rate of diabetes and diabetic vascular complications | 30 months

SECONDARY OUTCOMES:
Carotid intima-media thickness (IMT) | 30 months
Ankle brachial index (ABI) | 30 months
Urine albumin creatinine ratio (UACR) | 30 months
Estimated glomerular filtration rate (eGFR) | 30 months
Stage of diabetic retinopathy evaluated by fundus photograph | 30 months

CONTACTS AND LOCATIONS:
Overall Officials: Jiajun Zhao, MD,PhD, Study Chair — Shandong Provincial Hospital
Locations (1):
- Shandong Provincial Hospital, Jinan, Shandong, China